CLINICAL TRIAL: NCT02428478
Title: The Effect of Desipramine on Genioglossus Muscle Activity During Sleep in Healthy Control Subjects
Brief Title: Effect of Desipramine on Genioglossus Muscle Activity in Healthy Adults Study A
Acronym: DESOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Director, Sleep Disordered Breathing Lab, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BWH-2014P001033A
Record Dates: First submitted 2015-04-21; First posted 2015-04-28 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Desipramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desipramine First, Placebo Second (Active Comparator): Desipramine 200 mg administered 2 hours before normal sleep time on first study night, then a 1-week non-treatment period, then placebo-matching desipramine administered 2 hours before normal sleep time on second study night.
  Interventions: Drug: Desipramine; Drug: Placebo
- Placebo First, Desipramine Second (Active Comparator): Placebo-matching desipramine administered 2 hours before normal sleep time on first study night, then a 1-week non-treatment period, then desipramine administered 2 hours before normal sleep time on second study night.
  Interventions: Drug: Desipramine; Drug: Placebo

INTERVENTIONS:
Drug: Desipramine — 200 mg administered 2 hours before normal sleep time
  Other Names: Norpramine
Drug: Placebo — Placebo-matching desipramine administered 2 hours before normal sleep time

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal participants. Until recently, the search for medicines to activate pharyngeal muscles in sleeping humans has been discouraging. However, exciting new animal research has shown that drugs with noradrenergic and antimuscarinic effects can restore pharyngeal muscle activity to waking levels. In this protocol the investigators will test the effect of desipramine (a tricyclic antidepressant with strong noradrenergic and antimuscarinic effects) on genioglossus muscle activity (EMG GG) during sleep in healthy control participants.

DETAILED DESCRIPTION:
Two overnight sleep studies, a placebo night and a drug night, will be performed approximately one week apart in random order. The placebo or drug will be administered 2 hours before lights out. At least 15 minutes of quiet wakefulness will be recorded to quantify the participant's awake EMG GG activity. Participants will then sleep in the lateral position to minimize pharyngeal resistance similar to previous studies of this kind.

The same will be done for stable non-rapid eye movement (NREM) and rapid eye movement (REM) sleep (free of arousals and other artifacts). Both NREM and REM sleep will be analyzed, recognizing that REM is less frequent on these drugs.

During the second part of the night, the participants will be connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which can provide a wide range of pressures between 20 and -20 cm H2O in order to modify upper airway pressure and measure change in EMG GG as a function of epiglottic pressure (muscle responsiveness).

ELIGIBILITY:
Inclusion Criteria:

* Healthy control subjects

Exclusion Criteria:

* Cardiovascular disease other than well controlled hypertension
* Depression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wellman, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Taranto-Montemurro L, Edwards BA, Sands SA, Marques M, Eckert DJ, White DP, Wellman A. Desipramine Increases Genioglossus Activity and Reduces Upper Airway Collapsibility during Non-REM Sleep in Healthy Subjects. Am J Respir Crit Care Med. 2016 Oct 1;194(7):878-885. doi: 10.1164/rccm.201511-2172OC. PMID 26967681

RESULTS

PARTICIPANT FLOW:
Period: First Study Night
Arm/Group | Desipramine First, Placebo Second | Placebo First, Desipramine Second
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Second Study Night
Arm/Group | Desipramine First, Placebo Second | Placebo First, Desipramine Second
Started | 8 (1 participant did not return for the second study night) | 6 (2 participants did not return for the second study night)
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis. 4 participants were excluded: 3 due to intermittent electromyographic amplifier malfunction; and 1 did not sleep on both study nights.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27.5 [24.0 to 39.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Genioglossus Activity During Non-rapid Eye Movement (NREM) Sleep Measured as Percent of Wakefulness Activity
Description: Electromyography (EMG) was used to analyze genioglossus (GG) [EMG GG] muscle movement. EMG GG activity was recorded via standard needle electrodes inserted into the genioglossus (tongue) muscle. Activity of EMG GG was measured during wakefulness and sleep as % of maximum activation obtained pushing the tongue against closed teeth during wakefulness (GG%max). Sleep values were then expressed as %wakefulness value for tonic and phasic EMG GG activity. Tonic activity was defined as the lowest EMG GG value during expiration, phasic activity was calculated as the peak value during inspiration minus the tonic value.
Time Frame: 1 night
Population: All participants who were randomized, completed both study nights, and were included in the analysis. 4 participants were excluded: 3 due to intermittent electromyographic amplifier malfunction; and 1 did not sleep on both study nights.
Measure: Median (Inter-Quartile Range); unit: percent wakefulness
Groups:
- Desipramine: Desipramine 200 mg administered 2 hours before normal sleep time on the first study night or second study night.
- Placebo: Placebo-matching desipramine administered 2 hours before normal sleep time on the first study night or second study night.
Arm/Group | Desipramine | Placebo
Number analyzed (Participants) | 10 | 10
percent wakefulness
  Tonic | 96 [86 to 120] | 75 [50 to 92]
  Phasic | 84 [49 to 90] | 93 [74 to 106]
Statistical Analysis 1: Comparison: Desipramine vs Placebo; Tonic analysis; Test type: Other; p = 0.01, Wilcoxon Matched-Pairs Signed-Rank Test — P<0.05 considered statistically significant
Statistical Analysis 2: Comparison: Desipramine vs Placebo; Phasic analysis; Test type: Other; p = 0.38, Wilcoxon Matched-Pairs Signed-Rank Test — P<0.05 considered statistically significant

2. Secondary Outcome: Change in Pharyngeal Critical Collapsing Pressure (Pcrit) as a Measure of Upper Airway Collapsibility
Description: Participants were connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which provided a wide range of pressures between 20 and -20 cm H2O in order to modify upper airway pressure. Following a baseline recording period of 5 minutes, the CPAP level was reduced to varying suboptimal pressures. Change in Pcrit was used to determine the collapsibility of the upper airway under both passive and active conditions, and is expressed as Passive Pcrit: ventilation at a nasal pressure of 0 cm H2O when pharyngeal muscles are passive; Active Pcrit: ventilation at a nasal pressure of 0 cm H2O when pharyngeal muscles are active. Improved=more negative Pcrit.
Time Frame: 1 night
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cm H2O
Arm/Group | Desipramine | Placebo
Number analyzed (Participants) | 10 | 10
cm H2O
  Passive Pcrit | -10.0 [-15.2 to -5.8] | -8.1 [-10.4 to -6.3]
  Active Pcrit | -14.9 [-18.5 to -6.8] | -10.5 [-15.6 to -8.6]
Statistical Analysis 1: Comparison: Desipramine vs Placebo; Passive Pcrit; Test type: Other; p = 0.037, Wilcoxon Matched-Pairs Signed-Rank Test; Median Change = -0.6
Statistical Analysis 2: Comparison: Desipramine vs Placebo; Active Pcrit; Test type: Other; p > 0.5, Wilcoxon Matched-Pairs Signed-Rank Test

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of desipramine or placebo.
Arm/Group | Desipramine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes